CLINICAL TRIAL: NCT02325284
Title: Phase 1 Pilot Study of an Apparatus and Method to Objectively Measure Pain in Normal Healthy Adults.
Brief Title: Objective Measurement of Pain Using the Algometer
Status: Completed | Type: Observational
Sponsor: Julia Finkel (Other)
Collaborators: CoolCad Electronics, LLC; University of Maryland Engineering (Unknown)
Responsible Party: Sponsor-Investigator, Julia Finkel, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Other Study IDs: Algometer/Phase 1 pilot study
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy adults
  Interventions: Device: Pressure Algometer Testing

INTERVENTIONS:
Device: Pressure Algometer Testing
  Other Names: Wagner FPIX 50™ digital pressure algometer.

SUMMARY:
The development of tools for assessment and management of pain in newborns and children is a high priority and represents a significant unmet need. The inadequate treatment of pain and the overuse of analgesics can cause harmful consequences for neonates, infants, and children. To accomplish successful pain management in children one must first objectively assess pain. Thus, to address these critical issues with pain management, the Human Algometer and methods are under development by Drs. Julia Finkel and Zena Quezado, Pain Medicine Program (SZI) at Children's National Medical Center.

DETAILED DESCRIPTION:
It is generally recognized that pain assessment and management in newborns and children is an unmet need. According to the American Medical Association, "The pediatric population is at risk of inadequate pain management, with age-related factors affecting pain management in children. Children are often given minimal or no analgesia for procedures that would routinely be treated aggressively in adults. Although much is now known about pain management in children, it has not been widely or effectively translated into routine clinical practice."1 Although some clinically validated methods exist (e.g. CRIES, PPIP, Faces, etc.), no "gold standard" of pain assessment has been adopted in clinical practice. All are hindered by ambiguous behavioral correlates to the pain stimuli standards as well as the subjective variability inherent in both clinical and parent evaluators 2.

Other apparatus/methods for pain assessment suffer from similar shortcomings. For example, pain tolerance threshold (PTT) and current perception threshold (CPT) determinations both rely on verbal response from a patient. Those determinations are subjective and semi-quantitative and use electrical stimulation to directly excite both large and small diameter sensory nerve fibers. The CPT determination represents the minimum amount of a potentially noxious electrical stimulus that can be perceived, while the PTT determination represents the maximum amount of noxious electrical stimulation that can be tolerated when used as a clinical diagnostic tool. Thus, PTT depends on a subject's verbal response and requires patient exposure to aversive electrical stimulation, which causes both undesirable discomfort but also elicits the affective component of pain.

Therefore, the development of tools for assessment and management of pain in newborns and children is a high priority and represents a significant unmet medical need. Both inadequately treated pain or over administration of analgesics can have deleterious physiologic consequences for neonates, infants and children. While a number of methods are in use, no "gold standard" for pain assessment exists. (Anand 2007) To accomplish meaningful pain management in children one must first be able to objectively assess pain, particularly in patients who are (1) non-verbal (e.g. neonates, infants), (2) lacking understanding and adequate verbalization skills (e.g. young children, developmentally disabled individuals) and (3) patients with compromising neuropathic clinical presentations. To address these critical issues with pain management, the Human Algometer and method are under development by Drs. Finkel and Quezado from the Pain Medicine Program at the Sheikh Zayed Institute. In brief, this device integrates a neurospecific neurostimulation of sensory nerve fibers involved in pain response and near infra-red spectroscopy (NIRS) signal acquisition derived from pain related hemodynamic changes in the somatosensory cortex. The device has the ability to collect data on the NIRS response in the cerebral cortex to noxious stimulation provided by the neurostimulation component. Signal processing of data from this trial and subsequent trials will result in (1) the detection and optimization of a NIRS signal specific to increased neuronal blood flow over the somatosensory cortex (nociceptive response) and the frontal cortex (affective component). The individual neurostimulatory and NIRS signal acquisition components integrated into this novel device are based in part or whole on previously FDA approved devices from Neurotron, Inc. and Covidien plc (former Somanetics INVOS ™) respectively.

ELIGIBILITY:
Inclusion Criteria:

* the subject 18-65 years of age.
* the subject is a healthy adult with significant ongoing medical conditions
* the subject is willing to remain at the research site for the duration of the study session.
* the subject is willing and able to provide written informed consent to study participation.

Exclusion Criteria:

* the subject has consumed alcohol within the last 12 hours prior to testing
* subject has pain at the time of testing anywhere in the body

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Collection of data for signal processing that will generate the algorithms and data filters required to establish proof of concept for the novel technology. | one year
  The data collected and process from the human algometer will generate a specific NIRS nociceptive response to neurostimulation in the somatosensory cortex.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States